CLINICAL TRIAL: NCT06155266
Title: Combination of Leukocyte Cell Surface Biomarkers Measured by Cytometry, to Differentiate Bacterial From Viral Infections in Emergency Department: a Multicentric Cohort for the Validation of Diagnostic Performances
Acronym: CYTOBACT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231707
Record Dates: First submitted 2023-11-13; First posted 2023-12-04 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Bacterial and Viral Infections
Keywords: Bacterial infection; Viral infection; Flow cytometry; HLA-DR; CD64; MerTk; CD24; CX3CR1; CD169
MeSH Terms: conditions — Virus Diseases; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 2 additional whole blood samples of 6mL each will be taken — As part of the initial blood work-up, 2 additional samples of 6mL each of whole blood will be taken, to which 1mL of Cytodelics® Stabiliser will be added. The tubes will be mixed by inverting 10 to 15 times, incubated at +20°C for 10 minutes, then transported within 1 to 2 hours at 4°C by courier to the CRB at Pitié-Salpêtrière for aliquoting and freezing at -80°C . The expression level of cell surface markers will then be measured in series on an Aurora spectral cytometer, after frozen samples (1 to 2 aliquots) have been sent from the CRB-PSL to CIMI (INSERM U1135) at -80°C approximately once a month.
  Any remaining samples sent to CIMI will be destroyed once the analyses have been completed.

SUMMARY:
The characterization of the bacterial or viral etiology of an infectious event is required for both isolation decisions and rationale use of antibiotics. In emergency room (ER), the direct identification of the causal pathogen is rarely available in real-time. Alternative is the identification of the host-response to either a bacterial or viral infection. One of this host-response is the expression of peripheral leukocytes cell surface markers, measured by flow cytometry. Investigators and others have reported the high diagnostic performances of combination of cell surface biomarkers to differentiate bacterial from viral infection. The CYTOBACT study aims to confirm on a 500 patients multicentric cohort (200 having already been collected during another study: SEPTIMET), the best combinations for this diagnostic issue.

The study will be conducted in 3 emergency departments of APHP hospitals network in Paris, France. Patients with a suspicion of infection will be proposed to participate. No intervention will be introduced during the routine care in the (ER) which will be let at the discretion of the treating emergency physician. During the routine blood sampling in the ER, an additional 30 ml volume of whole blood will be collected, centrifugated, aliquoted and stored at -80°C for further measurement of the expression of a panel of cell surface markers. The participants will be followed up during their hospitalization (if any) and no longer than 28 days. Clinical data at admission, usual blood tests and all microbiological investigations performed during the hospital stay will be recorded into an electronic case record form (eCRF). Based on all those recorded data (excepted the results of flow cytometry for cell surface biomarkers) 2 independent adjudicators will qualify the infectious episode into bacterial,viral or no infection, and (if any) into infection, sepsis or septic shock (according to Sepsis 3.0 definitions).

Using different "machine learning" statistical tools, all the combination of the cell surface biomarkers will be tested to select those with the highest performance to differentiate bacterial from viral infection.

DETAILED DESCRIPTION:
Patients attending the ED of one of the participant centers for a suspicion of infection will be informed and asked to participate. After obtaining a non-opposition to participate, during the routine blood sampling performed in the ER, an additional volume of 30 ml of whole blood will be collected, aliquoted and stored at -80°C, comprising notably 12 ml of whole blood to which 1 ml of Cytodelics® Stabiliser will be added and incubated à room temperature for 10 mn before being aliquoted and stored at -80°C. The remaining whole blood will be collected on EDTA and Paxgen tubes, centrifugated, aliquoted and stored at -80°C for blood collection.

Clinical data at admission (past medical history, vital parameters, infectious source (if any), treatments delivered in the ER) will be recorded into an eCRF. The participants will be followed up until leaving the hospital and no longer than day-28. All the microbiology tests performed during the hospital stay will be also recorded into eCRF. The diagnostic performance of the combinations of cell surface markers will be evaluated against a diagnostic reference on the bacterial of viral qualification of each infectious event. This diagnostic reference will be established by an independant expert comitee after reviewing all the clinical, and biological data recorded (excepted the results of flow cytometry), in order to adjudicate between bacterial, viral or no infection, and among infected patients to classify into infection, sepsis or septic shock (sepsis 3.0).

After completing the recruitement of participants, a panel of cell surface markers will be measured by batch on a spectral cytometer, comprising notably the biomarkers of interest already published : HLA-DR, CD169 and CX3CR1 on monocytes, and MerTk, CD64 and CD24 on neutrophils.

The performances of the combinations of cell surface markers already identified in the littérature will be tested prioritarily. However, in order to refine the best combinations of biomarkers to discriminate bacterial from viral infection, machine learning algorithms like gradient boosting tree and support vector machine tools will be applied on the entire results of cell surface markers measured. The diagnostic performance will be evaluated calculating the sensitivity, specificity, area under the ROC curve of the biomarkers combinations selected.

ELIGIBILITY:
Inclusion Criteria:

* >18 year-old
* Attending one of the participant ED from Monday to Friday between 8:30 am to 3:00 pm
* With a suspicion of infection (defined by either a measured temperature above 38°C or any microbiology diagnostic test ordered during the routine care)
* Having blood sampling during routine care
* Informed and having expressed his/her non-opposition to participate

Exclusion Criteria:

* - Pregnancy
* No social insurance
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ER with a suspicion of infection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-08-14 (Estimated); Study Completion 2025-08-14 (Estimated)

PRIMARY OUTCOMES:
performances of cell surface markers combinations for diagnosis | through study completion, an average of 15 months
  area under the ROC curve of the different combinations of cell surface biomarkers for the diagnosis of bacterial or viral infection.

SECONDARY OUTCOMES:
performances of cell surface markers combinations for severity assesment | through study completion, an average of 15 months
  area under the ROC curve of the different combinations of cell surface biomarkers for the diagnosis of infetion, sepsis or septic shock
performances of cell surface markers combinations according to the age range of participants | through study completion, an average of 15 months
  area under the ROC curve of the different combinations of cell surface biomarkers in the subgroups 18 to 75 year-old and >75 year-old for the diagnosis and severity assesment

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service des urgences, Lariboisière, Paris
  - Service des urgences, Saint-Antoine, Paris
  - Service des urgences, Pitié Salpêtrière, Paris

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.